CLINICAL TRIAL: NCT05847205
Title: A Prospective, Single- Center, Phase IV, Interventional, Single Arm Trial for the Evaluation of Subcutaneous Recombinant Hirudin 15 mg (RB Variant) in Prophylaxis of Deep Vein Thrombosis (DVT) Post Major Orthopedic Operations
Brief Title: Study Evaluation of Recombinant Hirudin in Prophylaxis of Post-Operative Deep Vein Thrombosis
Acronym: Thromb-001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THRIVE-DVT
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Prophylaxis of Deep Vein Thrombosis
Keywords: r-Hirudin; Thrombexx; post-operative; prophylaxis; DVT

STUDY DESIGN:
Intervention Model Description: Prospective, Single arm, single-center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- r-Hirudin (Experimental): Patients will be treated with r-Hirudin (Thrombexx) for a total of 15 days beginning with 15 mg BID s.c starting 6 hours after surgery or upon adequate hemostasis and continued until end of study.
  Interventions: Drug: r-Hirudin

INTERVENTIONS:
Drug: r-Hirudin — 100 Patients will be treated with r-Hirudin (Thrombexx) for a total of 15 days beginning with 15 mg BID s.c starting 6 hours after surgery or upon adequate hemostasis and continued until end of study.
  Other Names: Thrombexx

SUMMARY:
This study aims to evaluate the efficacy and safety of r-Hirudin RB variant 15 mg in DVT prophylaxis post major orthopedic operations

DETAILED DESCRIPTION:
Prospective, Single arm, single-center

Phase IV

100 Patients will be treated with r-Hirudin (Thrombexx) for a total of 15 days beginning with 15 mg BID s.c starting 6 hours after surgery or upon adequate hemostasis and continued until end of study.

Patients undergoing major orthopedic operations

For Events of Deep Vein Thrombosis (DVT) within 15 days post-op.) All of the patients underwent Routine bilateral compression Doppler.

For Clinical PE (Pulmonary Embolism) Events from Day of surgery and During Hospitalization period or end of study

Clinical PE events PE (Pulmonary Embolism) events were confirmed by spiral CT.

For follow up:

APTT should be done before the first dose then after 4 & 8 hours of the first dose, then on days 1,8,15 post operatively.

Enrolment period: 3 months duration Follow-up duration: Follow-up per patient will be for a period of 15 days

Primary endpoint:

• Primary end points included new onset symptomatic thrombosis requiring medical or surgical intervention or death due to thrombosis defined as fatal PE, ischemic stroke, mesenteric thrombosis, or myocardial infarction

Secondary endpoint:

* The Secondary end point of major bleeding is defined as clinically evident hemorrhage associated with a hemoglobin decrease ≥ 2 g/dL that leads to a transfusion of ≥2 units of whole blood or packed red cells outside of the perioperative period (time from the start of the surgery or procedure and up to 12 hours after), or hemorrhage that is intracranial, retroperitoneal, or into a prosthetic joint.
* Recording serious adverse events (SAE)/ adverse events (AE) during the study duration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body Weight >60 kg
* Patients undergoing major orthopedic operations
* Patients ready to sign informed consent form (ICF)
* Patients should discontinue any agents that affect haemostasis prior to the study medication use unless strictly indicated. These agents include medications such as: anticoagulants, thrombolytics, non-steroidal anti- inflammatory agents (including Ketorolac tromethamine), preparations containing aspirin, systemic salicylates, ticlopidine, dextran 40, clopidogrel, other anti-platelet agents including glycoprotein IIb/IIIa antagonists or systemic glucocorticoids.

Exclusion Criteria:

* Significant bleeding injury such as solid organ laceration or intracranial bleed at discretion of attending physician
* Hypersensitivity to Hirudin or prior documented Allergy to its components
* Pregnant or breast feeding
* Hemorrhagic stroke in preceding 3 months
* abnormal baseline coagulation characterized by an INR >1.4, obtained at the discretion of the treating clinician
* Required therapeutic anticoagulation for atrial fibrillation, prior VTE, or mechanical heart valve
* Patients with a history of coagulation disorder
* Treatment with concomitant anti-platelet agent other than aspirin 326 mg or more daily (Platelet count< 100X109 /dl)
* Active bleeding
* Subjects with a life expectancy less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
new onset symptomatic thrombosis | up to 15 days post operative
  Primary end points included new onset symptomatic thrombosis requiring medical or surgical intervention or death due to thrombosis defined as fatal PE, ischemic stroke, mesenteric thrombosis, or myocardial infarction.

SECONDARY OUTCOMES:
Major bleeding | up to 12 hours after surgery
  The Secondary end point of major bleeding is defined as clinically evident hemorrhage associated with ahemoglobin decrease ≥ 2 g/dL that leads to a transfusion of ≥2 units of whole blood or packed red cells outside of the perioperative period
Adverse events | up to 15 days post operative
  Recording serious adverse events (SAE)/ adverse events (AE) during the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dr Soliman, PhD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT05847205/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT05847205/SAP_001.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT05847205/ICF_002.pdf